CLINICAL TRIAL: NCT05164926
Title: The Effects of the Use of St. John's Wort Oil With Massage in the Perineum on Episiotomy, Perineal Damage and Wound Healing
Brief Title: The Use of St. John's Wort Oil With Massage in the Perineum During Childbirth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Rahime Bedir Fındık, Associate Professor Dr, Ankara City Hospital Bilkent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent-MH-RBF-02
Record Dates: First submitted 2021-11-13; First posted 2021-12-21 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Perineal Injury
Keywords: perineal injury; perineal massage; St. John's Wort oil; Visual analogue scoring; episiotomy
MeSH Terms: interventions — Hypericum extract LI 160

STUDY DESIGN:
Intervention Model Description: two groups with St.John's Wort Oil control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group, whose perineum was massaged with St. John's Wort oil during labor (Experimental): St. John's Wort oil will be applied to this group during perineal massage during labor.
  Interventions: Other: perineal massage with St. John's Wort oil

INTERVENTIONS:
Other: perineal massage with St. John's Wort oil — perineal massage with St. John's Wort oil during labor

SUMMARY:
Perineal trauma, whether spontaneous or episiotomy, is a condition that affects the quality of life in primiparous women . In women who have experienced perineal trauma, problems such as dyspareunia, urinary and fecal incontinence, and delayed attachment of mother and baby occur in their later lives. Episiotomy, which is applied to reduce perineal trauma, is not recommended today, but it is still widely used.Different techniques such as perineal massage, hot compress, and Ritgen maneuver are applied to reduce perineal trauma. Perineal Massage can be applied together with oil. There are studies in which massage is applied together with oils.St. John's Wort (St. John's Wort) is a plant used in traditional practice in Turkish medicine against ulcers in the gastrointestinal tract, diabetes, jaundice, hepatic and biliary diseases. Antitumoral , antimicrobial , antiviral activities have been demonstrated. St. John's Wort oil can be used orally for dyspeptic complaints, and there is also a way to apply it through the skin. When applied for this purpose, it benefits from its facilitating feature of wound healing. It is useful in wound healing, myalgia and minor bruises, burn pain .

The investigators'aim in this study is to investigate the effects of perineal massage with St. John's Wort oil on episiotomy, perineal damage and wound healing.

DETAILED DESCRIPTION:
The study is a Prospective Cross-sectional Case Control study. 60 pregnant women who were admitted to the Delivery Room Clinic of the hospital for delivery and were in active labor and had a 6 cm gap of 70-80% in the examination were included in the study. High-risk pregnant women, pregnant women planned for cesarean delivery, and pregnant women with additional disease were excluded from the study. First of all, a patient follow-up form, which includes the demographic information of the pregnant women, examination and perineal length, ultrasound information including the estimated fetal weight of the baby, will be filled. 30 case group pregnant women will receive their consent following a detailed explanation. Then, perineal massage will be applied to the pregnant women who have reached full disclosure, which will last for 10 minutes in the 1st stage of labor, accompanied by centaury oil, to stretch the perineal muscles with the help of fingers. Also, the pregnant women who have reached full patency will be given a perineal massage until the head descends on the delivery table. Another 10-minute centaury oil massage will be applied.

The control group will consist of 30 pregnant women who were applied perineal massage without using centaury oil as a requirement of midwifery care service.

The rates of 3rd and 4th degree perineal damage will be recorded from the groups that received St. John's Wort oil after delivery and those who did not. The current cut-out size and depth and its localization will also be recorded. At the same time, the patient will be evaluated for VAS for postpartum perineal pain.

In the follow-up one week after discharge, the scar thickness and pelvic muscle strength assessment of the existing episioes and eruptions will be recorded. The presence of urinary or fecal incontinence will be recorded by asking.

The data will be saved in the IBM-SPSS program. When comparing the two groups, normally distributed data will be analyzed using the independent simple t test, and data not normally distributed will be analyzed using the Mann-Whitney U-Test. P value less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* normal pregnant women
* active labor during the examination
* pregnant woman who is likely to have a vaginal delivery

Exclusion Criteria:

.Pregnant women with risky pregnancies

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Presence of 3rd and 4th degree perineal damage | 5 minutes after birth
  The presence of 3rd and 4th degree perineal tears will be recorded by examination immediately after birth.
Visual Analogua Scale | 5 minutes after birth
  The scale has 0-10 points.As The point increases the pain score increases

SECONDARY OUTCOMES:
perineal muscle strength | postpartum at week 1
  Evaluation of perineal muscle strength by examination: The scale has 0-3 points. It is scored between a minimum of 0 and a maximum of 3.As the point increases the perineal muscle strenght score increases.
  0: no muscle strength
  1. weak muscle strength
  2. moderate muscle strength
  3. strong muscle strength
wound healing-wound color | postpartum at week 1
  Evaluation of wound color: The scale has 0-1 points.It is scored as 1 if the wound color is red and as zero (0) if it is not red.
wound healing-wound inflamation | postpartum at week 1
  Evaluation of wound inflamation: The scale has 0-1 points. It is scored as 1 if the wound is inflamed due to infection, and as zero (0) if it is not.
wound healing-wound heat | postpartum at week 1
  Evaluation of wound heat:The scale has 0-1 points.It is scored as 1 if there is an increase wound heat and zero (0) if there is none.

CONTACTS AND LOCATIONS:
Overall Officials: Rahime Bedir Findik, Dr, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Rahime Bedir Findik, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No